CLINICAL TRIAL: NCT05817409
Title: Predictive Factors for Treatment Success of Intrathecal Baclofen Therapy in Children With Cerebral Palsy - The Netherlands CP Register as a Unique Model for Practice Based, Long Term Data From Children With Cerebral Palsy.
Brief Title: Predictive Factors for Succes of ITB in CP
Status: Not yet recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Laura Bonouvrié, MD PhD, Amsterdam UMC, location VUmc
Other Study IDs: 2018.444
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cerebral Palsy; Intrathecal Baclofen
Keywords: cerebral palsy; intrathecal baclofen
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Intrathecal Baclofen Pump — intrathecal baclofen treatment
  Other Names: intrathecal baclofen treatment

SUMMARY:
For children with severe cerebral palsy (CP) in whom other options are insufficient, intrathecal baclofen (ITB) treatment could be an option. Literature provides some evidence for the effect of ITB, however we notice that not all children benefit equally. Furthermore long term effects of ITB in a prospective cohort of individuals with CP have not yet been described in literature. To improve selection for ITB physicians need to know which factors influence outcome on the long term. In order to accomplish these goals prospectively, real life data over a long period of time, and from a large cohort are needed.

The investigators will therefore conduct a prospective observational cohort study using the Netherlands CP register to collect data over a period of 4,5 years. The Netherlands CP register is an innovative register for data collection which was developed between 2016 and 2020 in a unique collaboration between children with CP, their parents, researchers and health care professionals.

All children and adolescents with CP, who start ITB treatment in the Netherlands under the age of 16, diagnosed with spastic or dyskinetic CP, are eligible for inclusion in the study.

The primary outcome measure is goal attainment scaling (GAS) in which achievement of individual goals can be quantified. Factors that potentially influence outcome including spasticity, dystonia, scoliosis and complications will be secondary outcome measures.

Measurements will be done before initiation of ITB, after 3 months, after 1 year and after 2 years.

Statistical analysis will include effect size Cohen's d for all outcome measures. To assess which factors are possibly associated with GAS T-score outcome at follow-up multiple regression analysis will be conducted.

DETAILED DESCRIPTION:
Background/rational:

Cerebral palsy (CP) is the most common cause of childhood disability with a prevalence of 2.11 per 1000 live births in high income countries. CP enfolds a group of developmental disorders of movement and posture, attributed to non-progressive disturbances which occurred in the developing foetal or infant brain.

An advanced treatment option for individuals with severe CP is Intrathecal Baclofen (ITB) treatment. This treatment can be considered when other options, such as oral medication, are insufficient or cause side effects. Previous studies have shown mostly low level evidence for the effect of ITB on spasticity in children with spastic CP. For children with dyskinetic CP, The Amsterdam UMC and Maastricht UMC previously conducted a randomized placebo-controlled trial, which provides evidence for the effect of ITB on attaining personal treatment goals after three months of ITB treatment. It was furthermore found that after one year of ITB treatment, personal treatment goals were at least partially achieved in 97% of children and adolescents.

Not all children show similar response to ITB: some benefit more than others in attaining treatment goals. The investigators previous research on the effect of ITB in children with dyskinetic CP, found that a higher level of dystonia prior to ITB and reduction of pain during ITB were associated, for a small part, with attainment of treatment goals. Sample size was not sufficient to look at specific factors associated with specific types of treatment goals. For example, goals on the level of personal care could be influenced by other factors than goals related to sitting or transfers.

Long-term effects of ITB in a prospective cohort of individuals with spastic and dyskinetic CP have not yet been described in literature. Furthermore, knowing which factors influence outcome on the long term, preferably related to specific types of treatment goals, can be used to inform and select children and adolescents with CP better before initiating ITB. In order to accomplish these goals prospectively, real life data over a long period of time, and from a large cohort are needed.

The Netherlands CP register is an innovative register for data collection which was developed between 2016 and 2020 in a unique collaboration between children with CP, their parents, researchers and health care professionals. The overall aim of the register is to provide personalized, value-based care for children with CP. In the Netherlands CP register, a follow-up registration program is combined with treatment registration.

Prospective data collection in the treatment registration will allow us to implement standardised assessment protocols in the two academic medical centres in the Netherlands where baclofen pump implantations are performed, the Amsterdam University Medical Center (Amsterdam UMC) in Amsterdam and Maastricht UMC (MUMC)in Maastricht.

Objectives:

The primary research question of this study is:

1. What is the short- (3 months), medium- (1 year) and long-term (2 years) effect of ITB in children with CP on personal treatment goals?

Secondary objectives are:

1. What is the association between the effect on personal treatment goals and on spasticity and/or dystonia?
2. Which factors are associated with treatment success of ITB in children with CP?

Study design A prospective observational study will be conducted in Amsterdam UMC and the MUMC using the Netherlands CP register to collect data over a period of 4,5 years. It is anticipated that in these centres 15 to 20 pumps will be implanted in children and adolescents annually. Over the total study period of 4,5 years, we aim to include a total of 67 to 90 children.

The Medical Ethics Review Committee (MEC) of the Amsterdam UMC, location VU University Medical Center (IRB00002991) has stated that the Medical Research Involving Human Subjects Act (WMO) does not apply to the study and that further official approval by the MEC is waived.

Participants Inclusion criteria

* All children with CP
* Who start ITB treatment in the Netherlands under the age of 16 Exclusion criteria
* no consent is given by the patient and/or caregiver for participation.

Subject follow up schedule In the investigators previous randomised controlled trial (the IDYS trial) on the effect of ITB in dyskinetic CP, we found that after three months of ITB most goals were, at least partially, attained. A study by Albright et al, additionally implies that dosage increases mostly in the first months, then shows some increase between 12 to 24 months and is fairly stable thereafter. Considering this information, data are collected and entered in the register at the following time points: before initiation of ITB, after 3 months, after 1 year, after 2 years. All centres participating in the register and performing ITB pump implantations enter data directly into the CP register. Data collection ceases if the patient dies, if ITB therapy is terminated, or once the patient transitions to adult services at the age of 18.

Outcome measures The primary outcome measure in this study is goal attainment scaling (GAS) in which achievement of individual goals can be quantified. Secondary outcome measures include: patient characteristics, treatment history, Range of motion, spasticity. Dystonia, scoliosis, selectivity, functional strength, gait analysis, questionnaires on activities and participation, treatment characteristics ITB including dosage, complications.

Statistical method/rationale A linear mixed-model analysis will be used to determine the development over time for the primary and secondary outcome measures, using time as a categorical variable. All analyses will be adjusted for possible covariates.

Effect size (ES) Cohen's d will be calculated for all outcome measures. Univariable linear regression analysis for each potential variable influencing outcome will be conducted. Factors showing a p-value of ≤0.20 are then selected for input in a final model in which a multiple regression analysis using backward stepwise selection will be performed to identify the predicting factors.

A p-value < 0.05 is considered statistically significant. Correction for multiple testing will be done by Holm correction of p-values.

ELIGIBILITY:
Inclusion Criteria:

* All children and adolescents diagnosed with CP,
* who start ITB treatment in the Netherlands under the age of 16,

Exclusion Criteria:

* no consent is given by the patient and/or caregiver for participation

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all patients with CP who start ITB under the age of 16 are eligible. They are recruited from the Amsterdam UMC or Maastricht UMC. Those are the only two centers in the Netherlands where ITB pump are implanted in children.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Goal Attainment Scaling (GAS) | 3 months, 1 year, 2 years
  Attainment of personal treatment goals are scored on a standardised scale where -2 is the baseline score and 0 is the goal. Scores can be given for deterioration (-3), improvement but not attainment (-1) and more (+1) or much more (+2) than goal achieved). change in these outcomes between the different time points is assessed.

SECONDARY OUTCOMES:
range of motion | baseline, 3 months, 1 year, 2 years
  range of motion of lower extremity joints
spasticity | baseline, 3 months, 1 year, 2 years
  Catch present or not
Barry-Albright-Dystonia Scale (BADS) | baseline, 3 months, 1 year, 2 years
  Dystonia is assessed in 8 body regions. A score of 0 to 4 can be given, where 0 represents no dystonia present, and 4 represents severe dystonia present.
Scoliosis | baseline, 3 months, 1 year, 2 years
  Cobb angle
Selective motor control testing | baseline, 3 months, 1 year, 2 years
  Selective control of movement of seperate joints is assessed for the hipflexors, knee-extensors and dorsiflexors of the foot. It is scored as normal, and if a patient can not move one joint seperatly from another joint, selectivity is scored as decreased (some selective control) or absent (no selective control at all)
Functional strength testing | baseline, 3 months, 1 year, 2 years
  Gross motor skills including squatting and toe walking are used to assess the functional strength of muscles. Normal strength testing is difficult in children with central nervous system motor disorders. Scores for the motor skills are: + child is able to execute motor skill, +/- child is able but with problems or incompletly, - child is not able to execute motor skill
walking pattern/gait analysis | baseline, 3 months, 1 year, 2 years
  walking pattern/gait analysis
Pediatric Evaluation of Disability Inventory (PEDI) | baseline, 3 months, 1 year, 2 years
  Questionnaire that assesses functional skilles, level of independence, and the extent of modifications required to perform functional activities in young children
Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) | baseline, 3 months, 1 year, 2 years
  The CPCHILD questionnaire is a validated measure of health-related quality of life for children with severe disabilities.
Pain severity on Visual Analogue Scale (pain VAS) | baseline, 3 months, 1 year, 2 years
  The severity of pain is score on a visual analogue scale (VAS) ranging from 0 to 10 where 0 represents no pain, and 10 the most excruciating pain possible
ITB pump details | 3 months
  Volume of ITB pump (20 ml or 40ml)
Catheter tip heigth | 3 months, 1 year, 2 years
  the height of the tip is assessed with insurgery X-ray. possibilities are: cervical, high thorecal (Th1-7), low thorecal (Th 8-12)
Catheter type | 3 months
  Different types of catheters are used. The specific cathter type (number provided by producer of pump) is used as an outcome measure
Complications | 3 months, 1 year, 2 years
  Complications related to ITB are noted.

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke Buizer, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Dutch CP register — https://cpregister.nl/